CLINICAL TRIAL: NCT06033846
Title: Efficacy and Safety of Adjunctive Minocycline in the Treatment of Autoimmune Encephalitis: Open-lable, Randomised, Proof of Concept Study
Brief Title: Efficacy and Safety of Adjunctive Minocycline in the Treatment of Autoimmune Encephalitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJLL-KY-20232121
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Encephalitis
Keywords: autoimmune encephalitis; minocycline
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Treatment group (Experimental): Drug: Minocyclin 200 mg oral minocycline for a total of 30 days
  Interventions: Drug: Minocycline
- Control group (No Intervention): first-line drugs for autoimmune encephalitis

INTERVENTIONS:
Drug: Minocycline — treatment with minocycline combined with first-line drugs for autoimmune encephalitis
  Other Names: minocycline hydrochloride
  Arms: Experimental: Treatment group

SUMMARY:
Autoimmune encephalitis (AE) is an immune-mediated brain disorder characterized by varied clinical manifestations that correlate with specific types of antibodies.Typical symptoms include acute behavioral changes, psychosis, seizures, memory deficits, dyskinesias, speech impairments, and autonomic and respiratory dysregulation.While the majority of patients respond well to immunotherapeutic agents, a significant proportion remains resistant to initial and secondary-line immunotherapies.Minocycline, a semisynthetic tetracycline, is notably used for the central nervous system due to its lipophilic characteristics and its capacity to penetrate the blood-brain barrier. While the primary neuroprotective focus of minocycline in the central nervous system remains unknown, the primary effects of minocycline include the inhibition of microglial activation, mitigation of apoptosis, and reduction in reactive oxygen species generation.Protective effect has been observed in hypoxic injury, ischemic stroke, amyotrophic lateral sclerosis, traumatic spinal cord injury, multiple sclerosis, Parkinson's disease, and Huntington's disease.Can minocycline offer a protective role in AE? Consequently, we proposed a randomized, controlled trial to investigate the efficacy of minocycline in AE.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of definite autoimmune encephalitis(Graus et al 2016.)
2. Age ≥ 18 years
3. Acute or subacute onset (rapid progression of less than 3 months)
4. Reasonable exclusion of alternative causes
5. Written informed consent

Exclusion Criteria:

1. Known allergy to tetracycline antibiotics.
2. Pregnant women.
3. Uncontrolled serious concomitant illness.
4. Known chronic kidney disease stages 3b-5.
5. Moderate liver disease (see Child-Pugh for Classification of Severity of Liver Disease).
6. history of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Montreal-Cognitive Assessment (MoCA)scores | 3 months
  the change in MoCA scores from baseline to 3 months

SECONDARY OUTCOMES:
modified rankin scale (mRS) scores | 1 month
  The proportion of patients achieving a ≥1-point or ≥2-point improvement in mRS scores at 1 month
MoCA scores | from baseline to months 1, 6, and 12
  change in MoCA scores from baseline to months 1, 6, and 12
mini-mental state examination (MMSE) scores | from baseline to months 1, 3, 6, and 12
  change in MoCA scores from baseline to months 1, 3, 6, and 12
Hamilton anxiety scale (HAMA) scores | from baseline to months 1, 3, 6, and 12
  changes in HAMA scores from baseline to months 1, 3, 6, and 12
Hamilton depression scale (HAMD) scores | from baseline to months 1, 3, 6, and 12
  changes in HAMA scores from baseline to months 1, 3, 6, and 12

OTHER OUTCOMES:
cerebrospinal fluid (CSF) levels of Soluble Triggering Receptor Expressed on Myeloid cells 2 (sTREM2) | from baseline to months 1, 3, 6, and 12.
  the change in CSF levels of sTREM2 levels from baseline to months 1, 3, 6, and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, China